CLINICAL TRIAL: NCT02554864
Title: Location of Injection of Local Anesthetics in the Adductor Canal Block: A Randomized Controlled Trial of the Effect on Postoperative Analgesia and Motor Power
Brief Title: Location of Injection of Local Anesthetics in the Adductor Canal Block
Acronym: LILAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-0046-B
Record Dates: First submitted 2015-09-09; First posted 2015-09-18 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Adductor Canal Block
MeSH Terms: interventions — Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adductor Canal Block- Injection -Site A (Active Comparator): AC Block-Injection (lidocaine 2% and ropivacaine 1%) Site A - after the sartorius muscle crosses over the femoral artery
  Interventions: Drug: lidocaine; Drug: ropivacaine
- Adductor Canal Block - Injection -Site B (Active Comparator): AC Block-Injection (lidocaine 2% and ropivacaine 1%) Site B - before the sartorius muscle crosses over the femoral artery
  Interventions: Drug: lidocaine; Drug: ropivacaine
- Adductor Canal Block -Injection -Site C (Active Comparator): AC Block-Injection (lidocaine 2% and ropivacaine 1%) Site C - as the sartorius muscle crosses over the femoral artery
  Interventions: Drug: lidocaine; Drug: ropivacaine

INTERVENTIONS:
Drug: lidocaine — Local anesthetic
  Other Names: Xylocaine
Drug: ropivacaine — Local anesthetic
  Other Names: Naropin

SUMMARY:
The adductor canal block (ACB) is the standard of care for analgesia after Anterior Cruciate Ligament (ACL) repair. ACB is performed by injecting local anesthetic (freezing) in the subsartorial canal in the thigh which is about 7-10cm long. Preliminary evidence suggests that different injection sites within the canal may produce different degrees of analgesia and quadriceps motor block. This trial seeks to determine the effects of various ACB injection sites on postoperative analgesia and motor power following ACL repair.

DETAILED DESCRIPTION:
Adductor canal block (ACB) is replacing femoral nerve block (FNB) as the peripheral nerve block of choice for knee surgery. The ACB aims to inject local anesthetics (LA) within the neurovascular sheath in the subsartorial adductor canal around the femoral nerve. The point where the sartorius muscle crosses over the femoral artery is generally the accepted site for performing ACB. Clinically, injecting LA in the adductor canal blocks the sensory innervation of the knee and thus offers pain relief that is similar to FNB while conserving motor power around the knee. While these benefits are desirable, the exact location for performing ACB that ensures these benefits, remains debatable. The subsartorial adductor canal itself is 7-10cm long and the anatomical location of the sensory and motor nerves that innervate the knee and its surrounding muscles in this canal may vary. This randomized controlled trial is designed to identify and refine the ACB technique by clinically determining the effects of various ACB injection locations on postoperative analgesia and quadriceps motor power following ACL repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients booked for anterior cruciate ligament surgery under general anesthesia
* English speaking
* BMI <38 kg/m2

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Allergy to local anesthetics
* Contraindication to regional anesthesia including coagulopathy or bleeding - diathesis
* Infection
* Nerve Injury at the site of the nerve block
* Malignancy at the site of the nerve block
* History of drug and/or alcohol dependence
* History of long term opioid intake or chronic pain disorder
* History of pre-existing neuropathy in the operative leg
* History of significant psychiatric conditions that may affect patient assessment
* Inability to understand the informed consent and demands of the study
* Allergy to any of the components of multi-modal analgesic regimen
* Revision ACL repair

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Cumulative 24 Hour Oral Morphine Equivalent Consumption | 24 hours
  Post-Operative Analgesia
Motor Power - Peak Force as measured by a dynamometer | 30 Minutes post Block
  Percentage decrease in quadriceps motor strength at 30 minutes following adductor canal block compare to baseline

SECONDARY OUTCOMES:
Opioid Consumption | During surgical procedure
  Intra-operative opioid consumption
Total opioids in Post Anesthetics (PAC) | Total length of time in PACU (total time in minutes from arrival in PACU to discharge to the Surgical Day Care is between 60-180 minutes
  Cumulative oral morphine equivalent consumption in PACU
Pain Scores - Questionnaire | 24 hours post block
  Area under the curve for rest pain scores plotted against time during the first 24 hours
Quality of Recovery (QoR-15) | 24 hours postoperatively
  Quality of recovery measured using the QoR-15 at 24 hours postoperatively
Patient Satisfaction - Questionnaire | 24 hours postoperatively
  Patient satisfaction with analgesia - NRS Pain Scale 0(no pain to 10(worst pain)
Hospital Discharge (Time to hospital discharge) | Same day as surgical procedure
  Time to hospital discharge
Nerve Block Complications | 24 hours postoperatively and 2 weeks postoperatively
  Presence/absence of nerve block complications during the first 24 hours postoperatively and 2 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University of Toronto, Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Mariano ER, Perlas A. Adductor canal block for total knee arthroplasty: the perfect recipe or just one ingredient? Anesthesiology. 2014 Mar;120(3):530-2. doi: 10.1097/ALN.0000000000000121. No abstract available. PMID 24534851
- [Background] Ilfeld BM, Hadzic A. Walking the tightrope after knee surgery: optimizing postoperative analgesia while minimizing quadriceps weakness. Anesthesiology. 2013 Feb;118(2):248-50. doi: 10.1097/ALN.0b013e318279fa3a. No abstract available. PMID 23241724
- [Background] Hanson NA, Derby RE, Auyong DB, Salinas FV, Delucca C, Nagy R, Yu Z, Slee AE. Ultrasound-guided adductor canal block for arthroscopic medial meniscectomy: a randomized, double-blind trial. Can J Anaesth. 2013 Sep;60(9):874-80. doi: 10.1007/s12630-013-9992-9. Epub 2013 Jul 3. PMID 23820968
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Background] Krombach J, Gray AT. Sonography for saphenous nerve block near the adductor canal. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):369-70. doi: 10.1016/j.rapm.2007.04.006. No abstract available. PMID 17720129
- [Background] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Tsui BC, Ozelsel T. Ultrasound-guided transsartorial perifemoral artery approach for saphenous nerve block. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):177-8; author reply 178. doi: 10.1097/AAP.0b013e31819a273e. No abstract available. PMID 19282716
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972
- [Background] Mariano ER, Kim TE, Wagner MJ, Funck N, Harrison TK, Walters T, Giori N, Woolson S, Ganaway T, Howard SK. A randomized comparison of proximal and distal ultrasound-guided adductor canal catheter insertion sites for knee arthroplasty. J Ultrasound Med. 2014 Sep;33(9):1653-62. doi: 10.7863/ultra.33.9.1653. PMID 25154949
- [Background] Bendtsen TF, Moriggl B, Chan V, Pedersen EM, Borglum J. Redefining the adductor canal block. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):442-3. doi: 10.1097/AAP.0000000000000119. No abstract available. PMID 25140514
- [Background] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Background] Chi J, Chiu B, Cao Y, Liu X, Wang J, Balu N, Yuan C, Xu J. Assessment of femoral artery atherosclerosis at the adductor canal using 3D black-blood MRI. Clin Radiol. 2013 Apr;68(4):e213-21. doi: 10.1016/j.crad.2012.12.002. Epub 2013 Jan 17. PMID 23332436
- [Background] Andersen HL, Andersen SL, Tranum-Jensen J. The spread of injectate during saphenous nerve block at the adductor canal: a cadaver study. Acta Anaesthesiol Scand. 2015 Feb;59(2):238-45. doi: 10.1111/aas.12451. Epub 2014 Dec 14. PMID 25496028
- [Background] Kapoor R, Adhikary SD, Siefring C, McQuillan PM. The saphenous nerve and its relationship to the nerve to the vastus medialis in and around the adductor canal: an anatomical study. Acta Anaesthesiol Scand. 2012 Mar;56(3):365-7. doi: 10.1111/j.1399-6576.2011.02645.x. PMID 22335278
- [Background] Head SJ, Leung RC, Hackman GP, Seib R, Rondi K, Schwarz SK. Ultrasound-guided saphenous nerve block--within versus distal to the adductor canal: a proof-of-principle randomized trial. Can J Anaesth. 2015 Jan;62(1):37-44. doi: 10.1007/s12630-014-0255-1. Epub 2014 Oct 22. PMID 25337966
- [Background] Shah NA, Jain NP. Is continuous adductor canal block better than continuous femoral nerve block after total knee arthroplasty? Effect on ambulation ability, early functional recovery and pain control: a randomized controlled trial. J Arthroplasty. 2014 Nov;29(11):2224-9. doi: 10.1016/j.arth.2014.06.010. Epub 2014 Jun 19. PMID 25041873
- [Background] Saranteas T, Anagnostis G, Paraskeuopoulos T, Koulalis D, Kokkalis Z, Nakou M, Anagnostopoulou S, Kostopanagiotou G. Anatomy and clinical implications of the ultrasound-guided subsartorial saphenous nerve block. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):399-402. doi: 10.1097/AAP.0b013e318220f172. PMID 21697687
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Espelund M, Fomsgaard JS, Haraszuk J, Mathiesen O, Dahl JB. Analgesic efficacy of ultrasound-guided adductor canal blockade after arthroscopic anterior cruciate ligament reconstruction: a randomised controlled trial. Eur J Anaesthesiol. 2013 Jul;30(7):422-8. doi: 10.1097/EJA.0b013e328360bdb9. PMID 23549123
- [Background] Kirkpatrick JD, Sites BD, Antonakakis JG. Preliminary experience with a new approach to performing an ultrasound-guided saphenous nerve block in the mid to proximal femur. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):222-3. doi: 10.1097/AAP.0b013e3181d24589. No abstract available. PMID 20216039